CLINICAL TRIAL: NCT01127633
Title: Continued Efficacy and Safety Monitoring of Solanezumab, an Anti-Amyloid β Antibody in Patients With Alzheimer's Disease
Brief Title: Continued Safety Monitoring of Solanezumab (LY2062430) in Alzheimer's Disease
Acronym: EXPEDITION EXT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Solanezumab did not meet the primary endpoint in study H8A-MC-LZAX.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11935; H8A-MC-LZAO (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-05-19; First posted 2010-05-21 (Estimated); Results first posted 2018-05-03 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-09

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — solanezumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Solanezumab (Experimental)
  Interventions: Drug: Solanezumab
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Solanezumab — 400 mg of solanezumab administered once every 4 weeks by intravenous infusion (IV) for up to 8 years.
  Other Names: LY2062430
  Arms: Solanezumab
Drug: Placebo — Participants were from feeder studies (LZAM or LZAN). Placebo administered intravenously every 4 weeks through Week 80.
  Arms: Placebo

SUMMARY:
This study is an open-label extension study in Alzheimer's patients who have completed participation in either solanezumab Clinical Trial H8A-MC-LZAM (NCT00905372) or H8A-MC-LZAN (NCT00904683).

ELIGIBILITY:
Inclusion Criteria:

* Meets National Institute of Neurological and Communicative Disorders and Stroke/Alzheimer's Disease and Related Disorders Association (NINCDS/ADRDA) criteria for probable Alzheimer's Disease
* Has completed participation in solanezumab Study LZAM or Study LZAN through 80 weeks
* Must continue to have a reliable caregiver who is in frequent contact with the patient for the entire study
* Must have good vein access to administer infusions
* Agrees not to participate in studies of any other investigational compounds for the duration of their participation in Study LZAO

Exclusion Criteria:

* Are currently enrolled in, or discontinued within the last 30 days from, a clinical trial involving an investigational drug or device or off-label use of a drug or device (other than the study drug/device used in this study), or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Meets LZAM or LZAN discontinuation criteria at the end of treatment in LZAM or LZAN study

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1457 (Actual)
Dates: Start 2010-12; Primary Completion 2014-07 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (147):
- United States (64):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Phoenix, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sun City, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tucson, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Little Rock, Arkansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Carson, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Laguna Hills, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lomita, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Los Angeles, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oxnard, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Diego, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Francisco, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santa Ana, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santa Monica, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Denver, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fairfield, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamden, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Haven, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Norwalk, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Newark, Delaware
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Washington D.C., District of Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boca Raton, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Myers, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hollywood, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miami Springs, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orange City, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orlando, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sunrise, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampa, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Atlanta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Canton, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Decatur, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lexington, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baltimore, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rockville, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Belmont, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Traverse City, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Creve Coeur, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Albuquerque, New Mexico
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Albany, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Amherst, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brooklyn, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Latham, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New York, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Staten Island, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Raleigh, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Winston-Salem, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beachwood, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toledo, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oklahoma City, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Eugene, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Portland, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., East Providence, Rhode Island
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charleston, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greer, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sioux Falls, South Dakota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salt Lake City, Utah
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bennington, Vermont
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Burlington, Vermont
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Norfolk, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Roanoke, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seattle, Washington
- Argentina (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buenos Aires
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ciudad Automona de Buenos Aire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Córdoba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mendoza
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rosario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santa Fe
- Australia (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gosford, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kogarah, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chermside, Queensland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toowoomba, Queensland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Box Hill, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Glen Iris, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heidelberg Heights, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Melbourne, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Subiaco, Western Australia
- Brazil (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Curitiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Itapira
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Porto Alegre
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rio de Janeiro
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., São Paulo
- Canada (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Medicine Hat, Alberta
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kelowna, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Penticton, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ottawa, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toronto, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greenfield Park, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sherbrooke, Quebec
- France (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paris
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rennes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Strasbourg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toulouse
- Germany (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hanover
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mannheim
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Munich
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Regensburg
- Italy (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baggiovara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Biella
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chieti
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Genova
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lido di Camaiore
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rome
- Japan (10):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aichi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ehime
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hiroshima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyōgo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kanagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kyoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shizuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo
- Poland (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bydgoszcz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gliwice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Katowice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Krakow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lublin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
- Russia (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chelyabinsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Petersburg
- South Korea (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Incheon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seongnam-si
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Suwon
- Spain (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Getafe
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Plasencia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Terrassa
- Sweden (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jönköping
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kalmar
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lund
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mölndal
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Umeå
- Taiwan (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guishan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Niaosong
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taipei
- United Kingdom (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Uckfield, E Susx
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Scotland, Glasgow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London, Greater London
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Camberwell, London

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who completed one of the feeder studies (Study LZAM (NCT00905372) or Study LZAN (NCT00904683)) were enrolled in this study.
Period: Overall Study
Arm/Group | Placebo | Solanezumab
Started | 723 | 734
Received at Least 1 Dose of Study Drug | 723 | 734
Completed | 70 | 61
Not Completed | 653 | 673
Not completed — Adverse Event | 74 | 73
Not completed — Death | 40 | 43
Not completed — Lost to Follow-up | 4 | 0
Not completed — Parent/Caregiver Decision | 246 | 228
Not completed — Physician Decision | 60 | 45
Not completed — Withdrawal by Subject | 57 | 72
Not completed — Sponsor Decision | 163 | 195
Not completed — Protocol Violation | 8 | 16
Not completed — Abnormal Lab/ECG Result | 0 | 1
Not completed — Not treated | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Solanezumab | Total
Number analyzed (Participants) | 723 | 734 | 1457
Age, Continuous [Mean (Standard Deviation); unit: Years] | 73.10 (8.004) | 72.96 (7.766) | 73.03 (7.883)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 406 | 415 | 821
  Male | 317 | 319 | 636
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 137 | 149 | 286
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 16 | 29
  White | 571 | 566 | 1137
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 41 | 40 | 81
  United States | 264 | 243 | 507
  Japan | 69 | 87 | 156
  United Kingdom | 17 | 18 | 35
  Spain | 15 | 22 | 37
  Russia | 13 | 15 | 28
  Canada | 38 | 40 | 78
  South Korea | 33 | 32 | 65
  Sweden | 21 | 15 | 36
  Taiwan | 26 | 23 | 49
  Poland | 18 | 25 | 43
  Brazil | 38 | 34 | 72
  Italy | 41 | 45 | 86
  Australia | 30 | 30 | 60
  France | 22 | 23 | 45
  Germany | 37 | 42 | 79

OUTCOME MEASURES:

1. Primary Outcome: Assess the Number of Participants With One or More Drug-Related Adverse Events (AEs) or Any Serious AEs (SAEs)
Description: The number of participants with 1 or more AEs assessed as related to the study drug and is summarized cumulatively. In addition, the number of participants with 1 or more serious AEs is summarized cumulatively. A serious AE is defined as an event that results in death, initial or prolonged hospitalization, is life-threatening, leads to persistent or significant disability/incapacity, is associated with congenital anomaly/birth defect, or is considered significant by the investigator for any other reason. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through Week 104
Population: All randomized participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | Solanezumab
Number analyzed (Participants) | 723 | 734
participants
  SAE | 308 | 299
  Other AE | 485 | 514

2. Secondary Outcome: Change From Baseline to 104-week Endpoint in Alzheimer's Disease Assessment Scale - Cognitive 14-Item Scale (ADAS-Cog14)
Description: ADAS-Cog14 is ADAS-Cog11 augmented with delayed free recall, digit cancellation, and maze completion measures. A score of 0 to 10 for delayed free recall and a conversion code of 0 to 5 for digit cancellation and maze completion provide total score ranges for this extended ADAS-Cog14 of 0 to 90. Higher scores indicate greater disease severity. Least Squares (LS) Mean was determined by mixed model repeated measures (MMRM) methodology with baseline, pooled investigator, treatment, visit, feeder visit 1 Mini-Mental State Examination (MMSE) status (mild/moderate), concomitant acetylcholinesterase inhibitors (AChEI)/Memantine use at baseline (yes/no), baseline age and treatment*visit.
Time Frame: Baseline, Week 104
Population: Feeder Intent-to-Treat Population: All randomized participants from feeder studies, who received at least one dose of study drug and had baseline & at least one post baseline observation for ADAS-Cog14.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Solanezumab
Number analyzed (Participants) | 409 | 451
Units on a scale | 17.58 (0.532) | 17.56 (0.517)
Statistical Analysis 1: Comparison: Placebo vs Solanezumab; Test type: Non-Inferiority or Equivalence — The noninferiority margin for this hypothesis was specified as 50% of the treatment difference observed at the end of the feeder study. If the lower limit of the confidence interval (CI) was greater than 0, the noninferiority criterion was met, indicating that at least 50% of the treatment difference observed at the end of the feeder studies was maintained at specified time points in the delayed-start period; p = 0.974, Mixed Models Analysis; Median Difference (Net) = -0.02, 95% CI 2-sided [-1.14 to 1.11]

3. Secondary Outcome: Change From Baseline to 104-week Endpoint in Alzheimer's Disease Cooperative Study - Activities of Daily Living Inventory (ADCS-ADL)
Description: ADCS-ADL is a 23-item inventory developed as a Rater-administered questionnaire answered by the participant's caregiver. It measures performance of basic and instrumental activities of daily living by participants. The total score ranges from 0 to 78, with lower scores indicating greater disease severity. LS Mean was determined by MMRM methodology with baseline, pooled investigator, treatment, visit, feeder visit 1 MMSE status (mild/moderate), concomitant AChEI/Memantine use at baseline (yes/no), baseline age and treatment*visit.
Time Frame: Baseline, Week 104
Population: Feeder Intent-to-Treat Population: All randomized participants from feeder studies, who received at least one dose of study drug and had baseline & at least one post baseline observation for ADCS-ADL.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Solanezumab
Number analyzed (Participants) | 420 | 456
Units on a scale | -26.77 (0.888) | -24.77 (0.871)

4. Secondary Outcome: Change From Baseline to 104-week Endpoint in Clinical Dementia Rating - Sum of Boxes (CDR-SB)
Description: CDR-SB is a semi-structured interview of participants and their caregivers. Participant's cognitive status is rated across 6 domains of functioning, including memory, orientation, judgment/problem solving, community affairs, home/hobbies, and personal care. Severity score assigned for each of 6 domains; Total score (SB) ranges from 0 to 18. Higher scores indicate greater disease severity. LS Mean was determined by MMRM methodology with baseline, pooled investigator, treatment, visit, feeder visit 1 MMSE status (mild/moderate), concomitant AChEI/Memantine use at baseline (yes/no), baseline age and treatment*visit.
Time Frame: Baseline, Week 104
Population: Feeder Intent-to-Treat Population: All randomized participants from feeder studies, who received at least one dose of study drug and had baseline & at least one post baseline observation for CDR-SB.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Solanezumab
Number analyzed (Participants) | 416 | 452
Units on a scale | 5.59 (0.174) | 5.27 (0.169)

5. Secondary Outcome: Change From Baseline to 104-week Endpoint in Neuropsychiatric Inventory (NPI)
Description: The NPI is a questionnaire administered to caregivers that quantifies behavioral changes in dementia. Each of the 12 behavioral domains the caregiver reports as present are scored for Frequency, scale: 1 (Occasionally) to 4 (Very Frequently), and Severity, scale: 1 (Mild) to 3 (Severe). If the domain is reported by the caregiver as 'Not Affected,' that domain is scored as 0. The individual domain scores are calculated by multiplying the frequency times the severity for each domain. NPI Total Score is calculated by adding the individual domain scores together for all 12 domains, with a scores range from 0 to 144. Lower scores indicated less severity and higher scores indicated a greater severity of neuropsychiatric disturbance. LS Mean was determined by MMRM methodology with baseline, pooled investigator, treatment, visit, concomitant AChEI/Memantine use at baseline (yes/no), baseline age and treatment*visit.
Time Frame: Baseline, Week 104
Population: Feeder Intent-to-Treat Population: All randomized participants from feeder studies, who received at least one dose of study drug and had baseline & at least one post baseline observation for NPI.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Solanezumab
Number analyzed (Participants) | 414 | 457
Units on a scale
  Mild Alzheimer's Disease: number analyzed (Participants) | 302 | 323
  Mild Alzheimer's Disease | 4.49 (0.788) | 5.41 (0.773)
  Moderate Alzheimer's Disease: number analyzed (Participants) | 112 | 134
  Moderate Alzheimer's Disease | 11.90 (1.517) | 8.10 (1.427)

6. Secondary Outcome: Change From Baseline to 104-week Endpoint in Resource Utilization in Dementia - Lite (RUD-Lite) Caregiver Hours
Description: The RUD-Lite is a caregiver-completed assessment designed to assess the amount of formal and informal resources used by participants and the primary caregiver. It is completed by the caregiver and compiles data on the following resources: length of time the caregiver spends giving care, assisting participants with basic activities of daily living (BADL: eating dressing, grooming, bathing); assisting participants with instrumental activities of daily living (IADLs: shopping, cooking, housekeeping, laundry, transportation, taking medication, managing finances), and providing supervision. Scores range from 0 to 24 hours. Higher values indicate greater resource use. LS Mean was determined by MMRM methodology with baseline, pooled investigator, treatment, visit, concomitant AChEI/Memantine use at baseline (yes/no), baseline age and treatment*visit.
Time Frame: Baseline, Week 104
Population: Feeder Intent-to-Treat Population: All randomized participants from feeder studies, who received at least one dose of study drug and had baseline & at least one post baseline observation for RUD-Lite.
Measure: Least Squares Mean (Standard Error); unit: hours per day (hr/day)
Arm/Group | Placebo | Solanezumab
Number analyzed (Participants) | 415 | 451
hours per day (hr/day)
  Mild Alzheimer's Disease-Basic ADL: number analyzed (Participants) | 302 | 319
  Mild Alzheimer's Disease-Basic ADL | 1.96 (0.184) | 1.21 (0.182)
  Mild Alzheimer's Disease-Instrumental ADL: number analyzed (Participants) | 303 | 319
  Mild Alzheimer's Disease-Instrumental ADL | 1.65 (0.207) | 1.05 (0.205)
  Mild Alzheimer's Disease-Supervision: number analyzed (Participants) | 303 | 319
  Mild Alzheimer's Disease-Supervision | 2.84 (0.368) | 2.59 (0.361)
  Moderate Alzheimer's Disease-Basic ADL: number analyzed (Participants) | 112 | 132
  Moderate Alzheimer's Disease-Basic ADL | 3.19 (0.461) | 3.54 (0.436)
  Moderate Alzheimer's Disease-Instrumental ADL: number analyzed (Participants) | 112 | 132
  Moderate Alzheimer's Disease-Instrumental ADL | 1.75 (0.461) | 1.72 (0.433)
  Moderate Alzheimer's Disease-Supervision: number analyzed (Participants) | 112 | 132
  Moderate Alzheimer's Disease-Supervision | 5.03 (0.693) | 4.47 (0.654)

7. Secondary Outcome: Change From Baseline to 104-week Endpoint in EuroQol 5-Dimensional Health-Related Quality of Life Scale Proxy Version (EQ-5D Proxy)
Description: EQ-5D (proxy version) is a generic, multidimensional, health-related, quality-of-life instrument assessing caregiver's impression of participants overall health state. Profile allows caregivers to rate participant's health state in 5 health domains: mobility, self-care, usual activities, pain/discomfort, and mood using a 3-level scale: 1 (no problem), 2 (some problems), and 3 (major problems). These attribute combinations are converted into a weighted Health-State Index Score according to the United States (US) population-based algorithm. EQ-5D US Population-Based Index Scores range from -0.11 to 1.0. A score of 1.0 indicated perfect health. The Overall Health State Index Score is caregiver-reported using a visual analogue scale marked 0 (worst imaginable health) to 100 (best imaginable health state). LS Mean was determined by MMRM methodology with baseline, pooled investigator, treatment, visit, concomitant AChEI/Memantine use at baseline (yes/no), baseline age and treatment*visit.
Time Frame: Baseline, Week 104
Population: Feeder Intent-to-Treat Population: All randomized participants from feeder studies, who received at least one dose of study drug and had baseline & at least one post baseline observation for EQ-5D Proxy.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Solanezumab
Number analyzed (Participants) | 414 | 453
Units on a scale
  Mild Alzheimer's Disease: number analyzed (Participants) | 303 | 320
  Mild Alzheimer's Disease | -0.07 (0.010) | -0.06 (0.009)
  Moderate Alzheimer's Disease: number analyzed (Participants) | 111 | 133
  Moderate Alzheimer's Disease | -0.16 (0.020) | -0.16 (0.019)

8. Secondary Outcome: Change From Baseline to 104-week Endpoint in Quality of Life in Alzheimer's Disease (QoL-AD)
Description: The QoL-AD (Caregiver Total Score) is a disease-specific measure of quality of life for an Alzheimer's Disease (AD) population administered to the participant's primary caregiver, who answers on behalf of the participant. The assessment consists of 13 items covering physical health, energy, mood, living situations, memory, family, marriage, friends, chores, fun, money, self and life as a whole. The assessment is scored on a 4-point Likert scale with scores ranging from 1 (poor) to 4 (excellent). QoL-AD Total Score is defined as the sum of the 13 items with a scores range from 13 to 52. Higher scores denote a better quality of life. LS Mean was determined by MMRM methodology with baseline, pooled investigator, treatment, visit, concomitant AChEI/Memantine use at baseline (yes/no), baseline age and treatment*visit.
Time Frame: Baseline, Week 104
Population: Feeder Intent-to-Treat Population: All randomized participants from feeder studies, who received at least one dose of study drug and had baseline & at least one post baseline observation for QoL-AD.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Solanezumab
Number analyzed (Participants) | 387 | 413
Units on a scale
  QLAD Self-Report Total Score-Mild Alzheimer's: number analyzed (Participants) | 273 | 283
  QLAD Self-Report Total Score-Mild Alzheimer's | -1.37 (0.331) | -0.98 (0.327)
  QLAD Caregiver Total Score-Mild Alzheimer's: number analyzed (Participants) | 284 | 299
  QLAD Caregiver Total Score-Mild Alzheimer's | -3.28 (0.350) | -3.63 (0.345)
  QLAD Self-Report Total Score-Moderate Alzheimer's: number analyzed (Participants) | 88 | 94
  QLAD Self-Report Total Score-Moderate Alzheimer's | -2.52 (0.605) | -2.34 (0.585)
  QLAD Caregiver Total Score-Moderate Alzheimer's: number analyzed (Participants) | 103 | 114
  QLAD Caregiver Total Score-Moderate Alzheimer's | -4.26 (0.573) | -3.14 (0.552)

9. Secondary Outcome: Change From Baseline to 104-week Endpoint in Mini-Mental State Examination (MMSE)
Description: The MMSE is an instrument used to assess a participant's cognitive function. The instrument is divided into 2 sections. The first section measures orientation, memory, and attention with scores ranging from 0 to 21 (lower scores indicate greater impairment). The second section tests the ability of the participant to name objects, follow verbal and written commands, write a sentence, and copy figures with scores ranging from 0 to 9 (lower scores indicate greater impairment). The range for MMSE Total Score is 0 to 30. Lower scores indicate more impairment. LS Mean was determined by MMRM methodology with baseline, pooled investigator, treatment, visit, concomitant AChEI/Memantine use at baseline (yes/no), baseline age and treatment*visit.
Time Frame: Baseline, Week 104
Population: Feeder Intent-to-Treat Population: All randomized participants from feeder studies, who received at least one dose of study drug and had baseline & at least one post baseline observation for MMSE.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Solanezumab
Number analyzed (Participants) | 412 | 446
Units on a scale | -8.08 (0.270) | -7.60 (0.263)

10. Secondary Outcome: Change From Baseline to 52-week Endpoint in Plasma Amyloid Beta (Aβ) Levels
Description: Concentration of the peptide Aβ 1-40 and Aβ 1-42 in plasma measured by immunoassay. The immunoassays for plasma Aβ 1-40 and Aβ 1-42 peptides were modified to render them tolerant to the presence of Solanezumab which would otherwise interfere with non-modified assays. LS Mean was determined by MMRM methodology with baseline, pooled investigator, treatment, visit, feeder visit 1 MMSE status (mild/moderate), concomitant AChEI/Memantine use at baseline (yes/no), baseline age and treatment*visit.
Time Frame: Baseline, Week 52
Population: All Feeder Intent-to-Treat Population: All randomized participants from feeder studies, who received at least one dose of study drug and had baseline & at least one post baseline observation for plasma Aβ 1-40 and Aβ 1-42.
Measure: Least Squares Mean (Standard Error); unit: picograms per milliliter (pg/mL)
Arm/Group | Placebo | Solanezumab
Number analyzed (Participants) | 515 | 532
picograms per milliliter (pg/mL)
  Aβ 1-40-Mild Alzheimer's Disease: number analyzed (Participants) | 358 | 357
  Aβ 1-40-Mild Alzheimer's Disease | 176412.04 (3718.292) | 173064.99 (3717.695)
  Aβ 1-42-Mild Alzheimer's Disease: number analyzed (Participants) | 356 | 356
  Aβ 1-42-Mild Alzheimer's Disease | 19854.92 (366.392) | 19723.48 (368.644)
  Aβ 1-40-Moderate Alzheimer's Disease: number analyzed (Participants) | 157 | 174
  Aβ 1-40-Moderate Alzheimer's Disease | 169356 (4627.8) | 169087 (4511.6)
  Aβ 1-42-Moderate Alzheimer's Disease: number analyzed (Participants) | 157 | 176
  Aβ 1-42-Moderate Alzheimer's Disease | 19237 (556.3) | 19552 (528.7)

11. Secondary Outcome: Change From Baseline to 104-week Endpoint in Volumetric Magnetic Resonance Imaging (vMRI)
Description: The vMRI assessment of right and left hippocampal volume is reported. LS Mean was determined by MMRM methodology with baseline, pooled investigator, treatment, visit, feeder visit 1 MMSE status (mild/moderate), concomitant AChEI/Memantine use at baseline (yes/no), baseline age and treatment*visit.
Time Frame: Baseline, Week 104
Population: Feeder Intent-to-Treat Population: All randomized participants from feeder studies, who received at least one dose of study drug and had baseline & at least one post baseline observation for vMRI.
Measure: Least Squares Mean (Standard Error); unit: Cubic millimeter (mm³)
Arm/Group | Placebo | Solanezumab
Number analyzed (Participants) | 310 | 325
Cubic millimeter (mm³)
  Right hippocampal volume-Mild Alzheimer's Disease: number analyzed (Participants) | 227 | 231
  Right hippocampal volume-Mild Alzheimer's Disease | -230.23 (8.232) | -230.07 (8.195)
  Left hippocampal volume-Mild Alzheimer's Disease: number analyzed (Participants) | 227 | 231
  Left hippocampal volume-Mild Alzheimer's Disease | -257.15 (8.153) | -244.00 (8.115)
  Right hippocampal volume-Moderate Alzheimer's: number analyzed (Participants) | 83 | 94
  Right hippocampal volume-Moderate Alzheimer's | -261.39 (11.796) | -256.52 (11.246)
  Left hippocampal volume-Moderate Alzheimer's: number analyzed (Participants) | 83 | 94
  Left hippocampal volume-Moderate Alzheimer's | -255.16 (11.466) | -253.29 (10.858)

12. Secondary Outcome: Change From Baseline to 104-week Endpoint in Alzheimer's Disease Assessment Scale - Cognitive Subscore 11-Item Scale (ADAS-Cog11)
Description: The cognitive subscale of the ADAS (ADAS Cog11) was used as a primary efficacy measure and consists of 11 items assessing areas of function most typically impaired in Alzheimer's disease: orientation, verbal memory, language, and praxis. The scale ranges from 0 to 70, with higher scores indicating greater disease severity. LS Mean was determined by MMRM methodology with baseline, pooled investigator, treatment, visit, feeder visit 1 MMSE status (mild/moderate), concomitant AChEI/Memantine use at baseline (yes/no), baseline age and treatment*visit.
Time Frame: Baseline, Week 104
Population: Feeder Intent-to-Treat Population: All randomized participants from feeder studies, who received at least one dose of study drug and had baseline & at least one post baseline observation for ADAS-Cog11.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Solanezumab
Number analyzed (Participants) | 375 | 409
units on a scale | 17.78 (0.595) | 17.38 (0.580)

13. Secondary Outcome: Mean Change From Baseline to Endpoint in Amyloid Imaging Parameters in Subjects With Mild Alzheimer's Disease
Description: Florbetapir PET imaging was used to test for change from baseline. The hypothesis that amyloid burden was reduced in participants between the treatment groups from the feeder studies was tested. The change from baseline to the postbaseline visit of the composite summary standard uptake value ratio of florbetapir F18 was calculated. The composite summary measure is an unweighted average of the 6 smaller regions (anterior cingulate, frontal medial orbital, parietal, posterior cingulate, precuneus, and temporal) normalized to whole cerebellum and to subject-specific white matter.
Time Frame: Baseline, Week 104
Population: Feeder Intent-to-Treat Population: All randomized participants with mild Alzheimer's Disease from feeder studies, who received at least one dose of study drug and had baseline & at least one post baseline observation for Amyloid Plaque Burden.
Measure: Mean (Standard Deviation); unit: Standard Uptake Value ratio (SUVr)
Arm/Group | Placebo | Solanezumab
Number analyzed (Participants) | 42 | 48
Standard Uptake Value ratio (SUVr) | 0.00 (0.131) | -0.01 (0.222)

ADVERSE EVENTS:
Description: There are gender specific adverse events, only occurring in male or female participants. The number of participants exposed has been adjusted accordingly.
Arm/Group | Placebo | Solanezumab
Serious Adverse Events (participants affected / at risk) | 308/723 | 299/734
Other Adverse Events (participants affected / at risk) | 485/723 | 514/734
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=723) | Solanezumab (N=734)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
Anaemia folate deficiency (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 4 (4) | 4 (5)
Angina pectoris (Cardiac disorders) | 2 (2) | 4 (5)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 5 (5) | 9 (9)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block (Cardiac disorders) | 2 (2) | 2 (2)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (3) | 2 (2)
Cardiac arrest (Cardiac disorders) | 5 (5) | 5 (5)
Cardiac failure (Cardiac disorders) | 2 (2) | 3 (3)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 6 (6) | 5 (5)
Cardiac perforation (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 2 (2) | 2 (2)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiovascular disorder (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 5 (5) | 4 (4)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 4 (4) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Myxoedema (Endocrine disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 3 (3) | 2 (3)
Glaucoma (Eye disorders) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1)
Strabismus (Eye disorders) | 1 (1) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colonic fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colonic pseudo-obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 0 (0)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticular fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Erosive oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 3 (3)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 2 (2) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 2 (2) | 4 (4)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 3 (3)
Jejunal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 5 (5) | 3 (3)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 2 (2)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal prolapse (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 3 (5) | 1 (1)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Subileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 3 (3)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abasia (General disorders) | 0 (0) | 1 (1)
Adverse drug reaction (General disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 5 (5) | 2 (2)
Catheter site haemorrhage (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 2 (2) | 1 (1)
Complication associated with device (General disorders) | 2 (2) | 0 (0)
Death (General disorders) | 4 (4) | 1 (1)
Drowning (General disorders) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 2 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (2) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 3 (3)
Sudden death (General disorders) | 3 (3) | 1 (1)
Bile duct obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 2 (2) | 2 (3)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Gallbladder polyp (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 2 (2)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 5 (5)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 7 (8)
Clostridium difficile colitis (Infections and infestations) | 2 (3) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 1 (1)
Colostomy infection (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 2 (2)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 4 (4) | 3 (3)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Escherichia sepsis (Infections and infestations) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Extradural abscess (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 3 (3)
Groin abscess (Infections and infestations) | 1 (1) | 0 (0)
Herpes simplex encephalitis (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (1)
Infected skin ulcer (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 2 (2) | 4 (4)
Labyrinthitis (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Mediastinitis (Infections and infestations) | 0 (0) | 1 (1)
Meningitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Orchitis (Infections and infestations) | 0/317 (0) | 1/319 (1)
Pericarditis tuberculous (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 27 (31) | 27 (31)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia pneumococcal (Infections and infestations) | 1 (1) | 1 (1)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 3 (3) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 3 (4) | 6 (6)
Septic shock (Infections and infestations) | 2 (2) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 16 (21) | 17 (19)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 3 (4) | 5 (7)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Bone contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (3)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 27 (27) | 23 (25)
Femoral neck fracture (Injury, poisoning and procedural complications) | 4 (4) | 13 (13)
Femur fracture (Injury, poisoning and procedural complications) | 11 (11) | 3 (3)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Flail chest (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fractured ischium (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Hip fracture (Injury, poisoning and procedural complications) | 8 (8) | 11 (12)
Humerus fracture (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 4 (4)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pubis fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pulmonary contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Rib fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal column injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 4 (4) | 5 (5)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Blood pressure increased (Investigations) | 1 (3) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Adult failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 7 (7) | 13 (15)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperammonaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperosmolar hyperglycaemic state (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypophagia (Metabolism and nutrition disorders) | 1 (1) | 1 (2)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 7 (7) | 13 (14)
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign soft tissue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Essential thrombocythaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Granular cell tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung carcinoma cell type unspecified stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3) | 0 (0)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/317 (0) | 1/319 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/406 (1) | 0/415 (0)
Altered state of consciousness (Nervous system disorders) | 2 (2) | 0 (0)
Brain stem haemorrhage (Nervous system disorders) | 2 (2) | 0 (0)
Brain stem infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haematoma (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 3 (3) | 1 (1)
Cerebral infarction (Nervous system disorders) | 3 (3) | 4 (4)
Cerebral microhaemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrospinal fluid leakage (Nervous system disorders) | 1 (3) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 3 (3)
Circadian rhythm sleep disorder (Nervous system disorders) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 0 (0) | 3 (3)
Coma (Nervous system disorders) | 0 (0) | 1 (1)
Complex partial seizures (Nervous system disorders) | 2 (2) | 0 (0)
Dementia alzheimer's type (Nervous system disorders) | 8 (8) | 5 (5)
Dementia with lewy bodies (Nervous system disorders) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Encephalopathy (Nervous system disorders) | 3 (4) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1) | 1 (1)
Generalised tonic-clonic seizure (Nervous system disorders) | 2 (2) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhagic cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial aneurysm (Nervous system disorders) | 1 (1) | 0 (0)
Intraventricular haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 6 (6) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 2 (2)
Loss of consciousness (Nervous system disorders) | 2 (2) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 1 (1)
Myoclonus (Nervous system disorders) | 1 (1) | 1 (1)
Normal pressure hydrocephalus (Nervous system disorders) | 2 (2) | 1 (1)
Presyncope (Nervous system disorders) | 2 (2) | 2 (2)
Seizure (Nervous system disorders) | 3 (3) | 11 (13)
Somnolence (Nervous system disorders) | 0 (0) | 2 (2)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 10 (10) | 15 (16)
Transient ischaemic attack (Nervous system disorders) | 3 (3) | 2 (2)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Vasogenic cerebral oedema (Nervous system disorders) | 1 (1) | 0 (0)
Abnormal behaviour (Psychiatric disorders) | 0 (0) | 1 (1)
Affective disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Aggression (Psychiatric disorders) | 2 (2) | 2 (7)
Agitation (Psychiatric disorders) | 11 (11) | 7 (7)
Alcohol abuse (Psychiatric disorders) | 0 (0) | 1 (1)
Behavioural and psychiatric symptoms of dementia (Psychiatric disorders) | 7 (10) | 3 (3)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 6 (6)
Delirium (Psychiatric disorders) | 5 (5) | 5 (5)
Delirium febrile (Psychiatric disorders) | 1 (1) | 0 (0)
Delusion (Psychiatric disorders) | 3 (3) | 2 (2)
Delusional perception (Psychiatric disorders) | 0 (0) | 1 (3)
Disorientation (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Irritability (Psychiatric disorders) | 3 (4) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 5 (5) | 2 (2)
Restlessness (Psychiatric disorders) | 2 (2) | 0 (0)
Suicidal behaviour (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 6 (6) | 2 (2)
Acute prerenal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Bladder tamponade (Renal and urinary disorders) | 0 (0) | 1 (1)
Calculus bladder (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 2 (2) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 3 (3) | 3 (3)
Acquired hydrocele (Reproductive system and breast disorders) | 0/317 (0) | 1/319 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2/317 (2) | 1/319 (1)
Cystocele (Reproductive system and breast disorders) | 1/406 (1) | 0/415 (0)
Prostatomegaly (Reproductive system and breast disorders) | 0/317 (0) | 1/319 (1)
Uterine prolapse (Reproductive system and breast disorders) | 1/406 (1) | 0/415 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 5 (6)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (6)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypersensitivity vasculitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Sebaceous gland disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Activities of daily living impaired (Social circumstances) | 1 (1) | 0 (0)
Cataract operation (Surgical and medical procedures) | 1 (2) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0)
Arterial thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 6 (7)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (2) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Shock (Vascular disorders) | 0 (0) | 1 (1)
Thromboangiitis obliterans (Vascular disorders) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=723) | Solanezumab (N=734)
Constipation (Gastrointestinal disorders) | 51 (56) | 64 (71)
Diarrhoea (Gastrointestinal disorders) | 58 (72) | 76 (105)
Vomiting (Gastrointestinal disorders) | 41 (51) | 51 (70)
Oedema peripheral (General disorders) | 31 (33) | 37 (38)
Bronchitis (Infections and infestations) | 32 (47) | 43 (56)
Nasopharyngitis (Infections and infestations) | 78 (129) | 88 (145)
Upper respiratory tract infection (Infections and infestations) | 59 (73) | 47 (61)
Urinary tract infection (Infections and infestations) | 98 (153) | 84 (161)
Contusion (Injury, poisoning and procedural complications) | 45 (62) | 58 (84)
Fall (Injury, poisoning and procedural complications) | 145 (222) | 136 (245)
Weight decreased (Investigations) | 48 (51) | 38 (40)
Decreased appetite (Metabolism and nutrition disorders) | 35 (39) | 37 (44)
Arthralgia (Musculoskeletal and connective tissue disorders) | 42 (51) | 33 (40)
Back pain (Musculoskeletal and connective tissue disorders) | 49 (54) | 67 (75)
Cerebral microhaemorrhage (Nervous system disorders) | 42 (47) | 56 (61)
Dizziness (Nervous system disorders) | 39 (43) | 43 (53)
Headache (Nervous system disorders) | 49 (65) | 46 (64)
Agitation (Psychiatric disorders) | 75 (83) | 64 (72)
Anxiety (Psychiatric disorders) | 56 (78) | 86 (114)
Insomnia (Psychiatric disorders) | 67 (70) | 74 (80)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 17/317 (17) | 9/319 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 50 (61) | 66 (74)
Hypertension (Vascular disorders) | 42 (43) | 36 (38)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days